CLINICAL TRIAL: NCT05668429
Title: A Phase 1, Open-Label, Single-Centre Study to Evaluate the Absorption, Distribution, Metabolism and Excretion (ADME) of Oral [14^C]-Ibrexafungerp in Healthy Male Subjects After Repeat Dosing
Brief Title: ADME Study of [14^C]-Ibrexafungerp in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCY-078-122
Record Dates: First submitted 2022-12-08; First posted 2022-12-29 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Fungal Disease
MeSH Terms: conditions — Mycoses | interventions — ibrexafungerp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose of [14^C]-Ibrexafungerp (Experimental): Each subject will receive a dose of [14C]-Ibrexafungerp at 12 h intervals for 7 doses in total.
  Interventions: Drug: Ibrexafungerp

INTERVENTIONS:
Drug: Ibrexafungerp — carbon-14 ([14^C])-Ibrexafungerp

SUMMARY:
This is a Phase 1, open-label, single center, non-randomized study to evaluate the absorption, distribution, metabolism and excretion (ADME) of an oral solution of radiolabeled Ibrexafungerp following repeat administration in healthy male subjects. All subjects will undergo preliminary screening procedures, will remain the clinical unit for approximately 26 days and will receive radiolabeled Ibrexafungerp, orally for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 30 to 65 years willing and able to sign and informed consent.

Exclusion Criteria:

* Clinically significant medical history or concurrent medical conditions included but not limited to infections, liver or kidney disease
* Use of certain concomitant medications
* History of smoking or alcohol abuse

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery | Day 26
  Mass balance recovery of total radioactivity in urine, faeces and all excreta (urine and faeces): cumulative recovery (CumAe) and cumulative recovery expressed as a percentage of the dose (Cum%Ae)
Metabolite identification in plasma, urine and faeces | Day 26
  Determination of primary metabolites using liquid chromatography-radio-detection
Area under the plasma concentration versus time curve (AUC) of Ibrexafungerp | Day1 and Day 4
  Area under the plasma concentration versus time curve (AUC) will be estimated where possible
Area under the plasma concentration versus time curve (AUC) of total radioactivity | Day 1 and Day 4
  Area under the plasma concentration versus time curve (AUC) of total radioactivity in blood where possible
Peak Plasma Concentration (Cmax) of Ibrexafungerp | Day 1 and Day 4
  Peak Plasma Concentration (Cmax) of Ibrexafungerp will be estimated

SECONDARY OUTCOMES:
Routes and rates of elimination of [14^C]-Ibrexafungerp | Day 26
  Determination of routes and rates of elimination of [14C]-Ibrexafungerp primarily by Ae total radioactivity for urine and faeces.
Distribution of total radioactivity into blood cells | Day 4
  Evaluation of whole blood plasma concentration ratios for total radioactivity
Safety of Ibrexafungerp | Day 4
  Number of participants with treatment-related adverse events as assessed by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Limited, Nottingham, United Kingdom